CLINICAL TRIAL: NCT06537180
Title: Gender-based Differences in the Outcome of the Treatment of Persistent Septic Shock With Hydrocortisone
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Other Study IDs: GBD-HYDRO
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Septic Shock
Keywords: Critical Care, Septic Shock, Hydrocortisone, Gender
MeSH Terms: conditions — Shock, Septic; Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The Female Group: Patients are categorized as females according to their apparent gender.
- The Male Group: Patients are categorized as males according to their apparent gender.

SUMMARY:
The aim of this study is to explore the gender-based differences in the outcomes of treatment with hydrocortisone in critically ill patients with persistent septic shock.

DETAILED DESCRIPTION:
Because of their pleiotropic effects, corticosteroids are widely used as adjunctive therapy in sepsis for their anti-inflammatory, metabolic, and immune-suppressing actions. Moreover, the treatment benefits of corticosteroids in terms of hemodynamics and organ functions for septic shock were established. Hydrocortisone reduces the duration of mechanical ventilation and critical care treatment and reduces the time needed for shock reversal. Hydrocortisone use at a daily dose of ≤400 mg for at least 3 days was associated with survival benefits.

Interestingly, corticosteroid treatment was reported to be more cost-effective in females than in males with septic shock, compared with placebo. This may be explained by the fact that sex hormones modulate the expression and sensitivity of glucocorticoid receptors differently, potentially influencing the body's response to cortisol. To the best of our knowledge, the data available on whether females and males may be more or less likely to acquire a better or worse prognosis of persistent septic shock when treated with hydrocortisone is sparse.

The aim of this study is to explore the gender-based differences in the outcomes of treatment with hydrocortisone in critically ill patients with persistent septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both sexes with persistent septic shock received hydrocortisone during their intensive care unit (ICU) stay.

Exclusion Criteria:

* Patients with incomplete data sets.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — According to apparent self-identified gender.
Study Population: Adult patients of both sexes with persistent septic shock received hydrocortisone during their intensive care unit (ICU) stay.
Sampling Method: Probability Sample
Enrollment: 621 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
28-day mortality | Day 28
  The rate of all-cause mortality after enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Alexandria University Hospitals, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moustafa HAM, Montasser M, Ahmed I, Mansy AEA, Habib T. Impact of sex on outcomes in septic shock patients treated with hydrocortisone. Sci Rep. 2025 Nov 29;15(1):42924. doi: 10.1038/s41598-025-28014-5. PMID 41318782